CLINICAL TRIAL: NCT01280656
Title: Retrospective Study to Evaluate the Impact of Using Interferon (Pegylated or Not) in the Treatment of Patients With Chronic Hepatitis C in Brazil (DECISION)
Brief Title: A Retrospective Study to Assess the Impact of the Use of Interferon in Patients With Chronic Hepatitis C (DECISION)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22995
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Results first posted 2016-09-26 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Conventional Interferon Plus Ribavirin: Eligible participants who will receive conventional interferon plus ribavirin for Chronic Hepatitis C (CHC) according to the standard of care and aligned with the local prescription instructions will be observed during treatment period (48 weeks) and follow up period (24 weeks).
  Interventions: Drug: Conventional Interferon; Drug: Ribavirin
- Peginterferon Alfa-2a Plus Ribavirin: Eligible participants who will receive peginterferon alfa-2a plus ribavirin for CHC according to the standard of care and aligned with the local prescription instructions will be observed during treatment period (48 weeks) and follow up period (24 weeks).
  Interventions: Drug: Peginterferon Alfa-2a; Drug: Ribavirin
- Peginterferon Alfa-2b Plus Ribavirin: Eligible participants who will receive peginterferon alfa-2b plus ribavirin for CHC according to the standard of care and aligned with the local prescription instructions will be observed during treatment period (48 weeks) and follow up period (24 weeks).
  Interventions: Drug: Peginterferon Alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Drug: Conventional Interferon — Conventional interferon according to the standard of care and aligned with the local prescription instructions
  Groups: Conventional Interferon Plus Ribavirin
Drug: Peginterferon Alfa-2a — Peginterferon alfa-2a according to the standard of care and aligned with the local prescription instructions
  Groups: Peginterferon Alfa-2a Plus Ribavirin
Drug: Peginterferon Alfa-2b — Peginterferon alfa-2b according to the standard of care and aligned with the local prescription instructions
  Groups: Peginterferon Alfa-2b Plus Ribavirin
Drug: Ribavirin — Ribavirin according to the standard of care and aligned with the local prescription instructions

SUMMARY:
This retrospective study will assess the sustained virologic response and the safety of two different interferons (pegylated or conventional) in patients with chronic hepatitis C. Data will be collected for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years and <70 years of age
* Diagnosis of hepatitis C
* Assessment of viral load prior to treatment (mandatory for genotype 1 only)
* Liver biopsy
* Co-morbidities data
* Use of interferon (pegylated or conventional) and ribavirin to treat hepatitis C infection genotype 2 and 3 and pegylated interferon plus ribavirin to treat hepatitis C infection genotype 1
* Above mentioned treatment started between 01-Sep-2007 and 31-Aug-2008

Exclusion Criteria:

* Co-infection with human immunodeficiency virus
* Co-infection with hepatitis B virus
* Presence of hepatocarcinoma
* Patients submitted to hemodialysis
* Organ transplant patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis C patients that received interferon (pegylated or conventional) during the period stipulated (from 01-Sep-2007 to 31-Aug-2008)
Sampling Method: Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- Brazil (27):
  - Rio Branco, Acre
  - Manaus, Amazonas
  - Vitória, Espírito Santo
  - Salvador, Estado de Bahia
  - Goiânia, Goiás
  - São Luís, Maranhão
  - Campo Grande - MS, Mato Grosso do Sul
  - Pouso Alegre, Minas Gerais
  - Uberaba, Minas Gerais
  - Curitiba, Paraná
  - Belém, Pará
  - Recife, Pernambuco
  - Niterói, Rio de Janeiro
  - Nova Iguaçu, Rio de Janeiro
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Rio Grande, Rio Grande do Sul
  - Porto Velho, Rondônia
  - Sao Jose Do Rio Preto, Santa Catarina
  - Aracaju, Sergipe
  - Botucatu, São Paulo
  - Campinas, São Paulo
  - Ribeirão Preto, São Paulo
  - Santo André, São Paulo
  - Santos, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 660 participants were enrolled from 39 centers in Brazil. The study was conducted from January 2010 to June 2013.
Groups:
- Conventional Interferon Plus Ribavirin: Eligible participants who received conventional interferon plus ribavirin for Chronic Hepatitis C (CHC) according to the standard of care and aligned with the local prescription instructions were observed during treatment period (48 weeks) and follow up period (24 weeks).
- Peginterferon Alfa-2a Plus Ribavirin: Eligible participants who received peginterferon alfa-2a plus ribavirin for CHC according to the standard of care and aligned with the local prescription instructions were observed during treatment period (48 weeks) and follow up period (24 weeks).
- Peginterferon Alfa-2b Plus Ribavirin: Eligible participants who received peginterferon alfa-2b plus ribavirin for CHC according to the standard of care and aligned with the local prescription instructions were observed during treatment period (48 weeks) and follow up period (24 weeks).
Period: Overall Study
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Started | 62 | 312 | 286
Completed | 59 | 265 | 223
Not Completed | 3 | 47 | 63
Not completed — Adverse Event | 1 | 14 | 13
Not completed — Lack of Efficacy | 1 | 22 | 38
Not completed — Treatment shortening (RGT) | 0 | 4 | 5
Not completed — Other | 1 | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Conventional Interferon Plus Ribavirin: Eligible participants who received conventional interferon plus ribavirin for CHC according to the standard of care and aligned with the local prescription instructions were observed during treatment period (48 weeks) and follow up period (24 weeks).
- Total: Total of all reporting groups
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin | Total
Number analyzed (Participants) | 62 | 312 | 286 | 660
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (8.6) | 49.2 (10.7) | 49.5 (9.5) | 49.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 188 | 147 | 357
  Male | 40 | 124 | 139 | 303

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at 12 Weeks After End of Treatment
Description: Sustained virological response (SVR) was defined as virological response at 12 weeks after end of treatment (EOT). Virologic response was either defined as having undetectable (that is, no hepatitis C virus Ribonucleic acid [HCV RNA] was detected in the participants' plasma samples) or less than 50 international units/milliliter (IU/mL) HCV RNA (that is, the participants' plasma samples contained traces of HCV RNA at a concentration below the limit of quantification of the viral load assay or no HCV RNA was detected in the samples). EOT= Week 48. Participants who did not have viral load assessment at Week 12 were considered treatment failures, except in the specific case where the lack of assessment was not due to treatment shortening in function of response guided therapy.
Time Frame: At Week 60
Population: The intent-to-treat (ITT) population consisted of participants who fulfilled all inclusion/ exclusion criteria. The analysis was performed in participants with virologic response at EOT in each group (16, 126, and 101 respectively).
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 16 | 126 | 101
percentage of participants | 0 | 7.1 | 20.8
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin vs Peginterferon Alfa-2b Plus Ribavirin; Test type: Superiority or Other; p = 0.003, Chi-squared

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 24 Weeks After End of Treatment
Description: SVR was defined as virological response at 24 weeks after EOT, EOT= Week 48. Virologic response was either defined as having undetectable (that is, no hepatitis C virus Ribonucleic acid [HCV RNA] was detected in the participants' plasma samples) or less than 50 IU/mL HCV RNA (that is, the participants' plasma samples contained traces of HCV RNA at a concentration below the limit of quantification of the viral load assay or no HCV RNA was detected in the samples). Participants who did not have viral load assessment at Week 12 were considered treatment failures, except in the specific case where the lack of assessment was not due to treatment shortening in function of response guided therapy.
Time Frame: At Week 72
Population: The ITT population consisted of participants who fulfilled all inclusion/ exclusion criteria. The analysis was performed in participants with virologic response at EOT in each group (16, 126, and 101 respectively).
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 16 | 126 | 101
percentage of participants | 62.5 | 74.6 | 72.3
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin vs Peginterferon Alfa-2b Plus Ribavirin; Test type: Superiority or Other; p = 0.693, Chi-squared

3. Secondary Outcome: Number of Participants With Interferon Dose Reduction Rates in Function of the Interferon Type Being Used
Description: The number of participants with Interferon dose reduction rates in function of the interferon type being used are reported
Time Frame: At Week 24
Population: The ITT population consisted of participants who fulfilled all inclusion/ exclusion criteria. The analysis was performed in the participants who were available for interferon dose reduction rates in each group (56, 302, and 280 respectively).
Measure: Number; unit: participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 56 | 302 | 280
participants | 1 | 9 | 29

4. Secondary Outcome: Percentage of Participants With Early Virologic Response at Week 12
Description: An early virologic response (EVR) was defined as a HCV-RNA decrease of at least two logarithmic scales (2 Log) or 100 times the pretreatment value or non-detection at Week 12 of treatment period.
Time Frame: At Week 12
Population: The ITT population consisted of participants who fulfilled all inclusion/ exclusion criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 62 | 312 | 286
percentage of participants | 14.5 | 37.2 | 35.0
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin vs Peginterferon Alfa-2b Plus Ribavirin; Test type: Superiority or Other; p = 0.573, Chi-squared

5. Secondary Outcome: Percentage of Participants With Sustained Virologic Response Treated at Interferon Application Centers and Treated at Home
Description: The percentage of participants with SVR-12 and SVR-24 treated at interferon application centers (IAC) and treated at home are presented.
Time Frame: At Week 60 (SVR 12) and Week 72 (SVR 24)
Population: The ITT population consisted of participants who fulfilled all inclusion/ exclusion criteria. The analysis was performed in participants with virologic response at EOT in each group excluding participants treated at an unknown location (2/16, 5/126, and 9/101 respectively).
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 14 | 121 | 92
percentage of participants
  SVR-12, treated at IAC (n=0, 40, 35) | NA — No participants were available for analysis in this arm. | 5.0 | 2.9
  SVR-12, treated at home (n=14, 81, 57) | 0 | 8.6 | 33.3
  SVR-24, treated at IAC (n=0, 40, 35) | NA — No participants were available for analysis in this arm. | 80.0 | 77.1
  SVR-24, treated at home (n=14, 81, 57) | 64.3 | 75.3 | 68.4

6. Secondary Outcome: Percentage of Participants Who Were Treated at Interferon Application Centers and at Home and Discontinued Treatment
Description: The percentage of participants who were treated at interferon application centers and at home and who discontinued treatment is presented. Participants who did not have viral load assessment at Week 12 were considered treatment failures, except in the specific case where the lack of assessment was not due to treatment shortening in function of response guided therapy.
Time Frame: Up to Week 48
Population: The ITT population consisted of participants who fulfilled all inclusion/ exclusion criteria. The analysis excluded participants treated at an unknown location (7/62, 10/312, and 23/286 respectively)
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 55 | 302 | 263
percentage of participants
  At the site (n=0,98,126) | NA — No participants were available for analysis in this arm. | 17.4 | 17.5
  At home (n=55,204,137) | 5.5 | 11.8 | 21.9
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin vs Peginterferon Alfa-2b Plus Ribavirin; Mean at the site; Test type: Superiority or Other; p = 0.982, Chi-squared
Statistical Analysis 2: Comparison: Peginterferon Alfa-2a Plus Ribavirin vs Peginterferon Alfa-2b Plus Ribavirin; Mean at home; Test type: Superiority or Other; p = 0.012, Chi-squared

7. Secondary Outcome: Mean Percentage Reduction of Hemoglobin in Treatment Responders and Treatment Non-Responders
Description: The average percentage reduction of hemoglobin (Hb) in treatment responders and treatment non-responders between the conventional group, peginterferon alfa-2a plus and peginterferon alfa-2b is presented. Participants with undetectable HCV RNA at specified time points (Weeks 4/12/18/24/48) were considered as treatment responders. Participants with positive viral load (detectable HCV RNA) at end of treatment regardless of the treatment duration were considered as treatment non-responders.
Time Frame: Up to Week 72
Population: The ITT population consisted of participants who fulfilled all inclusion/ exclusion criteria. Treatment responders and non-responders for whom data was available were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: mean percentage reduction of hemoglobin
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 10 | 73 | 63
mean percentage reduction of hemoglobin
  Responders (n=0,19,15) | NA (NA) — No participants were available for analysis in this arm. | 14.4 (8.5) | 15.8 (10.3)
  Non-responders (n=10,54,48) | 18.3 (9.5) | 9.8 (27.7) | 12.6 (11.1)
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin; Responders vs Non-responders; Test type: Superiority or Other; p = 0.476, t-test, 2 sided
Statistical Analysis 2: Comparison: Peginterferon Alfa-2b Plus Ribavirin; Responders vs Non-Responders; Test type: Superiority or Other; p = 0.320, t-test, 2 sided

8. Secondary Outcome: Percentage of Participants With Rapid Virologic Response at Week 4
Description: Rapid virologic response was defined as qualitative or quantitative HCV-RNA (viral load) undetectable (below the lower limit of detection) at Week 4 of treatment period.
Time Frame: At Week 4
Population: The ITT population consisted of participants who fulfilled all inclusion/ exclusion criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 62 | 312 | 286
percentage of participants | 6.5 | 21.2 | 20.3
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin vs Peginterferon Alfa-2b Plus Ribavirin; Test type: Superiority or Other; p = 0.792, Chi-squared

9. Secondary Outcome: Percentage of Participants With Virologic Response at End of Treatment
Description: Virologic response at EOT was defined as undetectable HCV-RNA at EOT (regardless in which week treatment was concluded). EOT = Week 48.
Time Frame: At Week 48
Population: The ITT population consisted of participants who fulfilled all inclusion/ exclusion criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 62 | 312 | 286
percentage of participants | 25.8 | 40.4 | 35.3
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin vs Peginterferon Alfa-2b Plus Ribavirin; Test type: Superiority or Other; p = 0.202, Chi-squared

10. Secondary Outcome: Percentage of Participants With Virologic Relapse up to Week 72
Description: Virologic relapse was defined as undetectable HCV-RNA at end of treatment and detectable HCV-RNA at the last follow-up assessment available. If the participant was a responder at end of treatment and was not submitted to any viral load assessment during the follow-up period, he was considered a relapser.
Time Frame: Up to Week 72
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 16 | 126 | 101
percentage of participants | 37.5 | 22.2 | 22.8
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin vs Peginterferon Alfa-2b Plus Ribavirin; Test type: Superiority or Other; p = 0.921, Chi-squared

11. Secondary Outcome: Percentage of Participants With Null Response or No Responder at End of Treatment
Description: Null response or no responders were defined as those participants presenting positive viral load at EOT (regardless of the treatment duration). EOT= Week 48.
Time Frame: At Week 48
Population: The ITT population consisted of participants who fulfilled all inclusion/ exclusion criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 62 | 312 | 286
percentage of participants | 74.2 | 59.6 | 64.7
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin vs Peginterferon Alfa-2b Plus Ribavirin; Test type: Superiority or Other; p = 0.202, Chi-squared

12. Secondary Outcome: Percentage of Participants Who Discontinued Treatment Due to Adverse Events
Description: The percentage of participants with treatment discontinuation rates due to adverse events (AE) between conventional group, peginterferon alfa-2a and peginterferon alfa-2b is presented.
Time Frame: Up to Week 48
Population: The ITT population consisted of participants who fulfilled all inclusion/ exclusion criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 62 | 312 | 286
percentage of participants | 1.6 | 4.5 | 4.6
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin vs Peginterferon Alfa-2b Plus Ribavirin; Total; Test type: Superiority or Other; p = 0.973, Chi-squared

13. Secondary Outcome: Number of Participants With Any Adverse Events and Any Serious Adverse Events
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event in the investigator's judgment or requires intervention to prevent one or other of these outcomes.
Time Frame: Up to Week 72
Population: The ITT population consisted of participants who fulfilled all inclusion/ exclusion criteria.
Measure: Number; unit: participants
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Number analyzed (Participants) | 62 | 312 | 286
participants
  any AE | 57 | 285 | 264
  any SAE | 2 | 15 | 9

ADVERSE EVENTS:
Time Frame: Up to Week 72
Description: Serious adverse events and non-serious adverse events are reported in ITT population set.
Groups:
- Conventional Interferon Plus Ribavirin: Eligible participants who received conventional interferon plus ribavirin for CHC according to the standard of care and aligned with the local prescription instructions were retrospectively assessed up to a minimum of 12 weeks after the end of therapy.
- Peginterferon Alfa-2a Plus Ribavirin: Eligible participants who received peginterferon alfa-2a plus ribavirin for CHC according to the standard of care and aligned with the local prescription instructions were retrospectively assessed up to a minimum of 12 weeks after the end of therapy
- Peginterferon Alfa-2b Plus Ribavirin: Eligible participants who received peginterferon alfa-2b plus ribavirin for CHC according to the standard of care and aligned with the local prescription instructions were retrospectively assessed up to a minimum of 12 weeks after the end of therapy.
Arm/Group | Conventional Interferon Plus Ribavirin | Peginterferon Alfa-2a Plus Ribavirin | Peginterferon Alfa-2b Plus Ribavirin
Serious Adverse Events (participants affected / at risk) | 2/62 | 15/312 | 9/286
Other Adverse Events (participants affected / at risk) | 55/62 | 275/312 | 262/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional Interferon Plus Ribavirin (N=62) | Peginterferon Alfa-2a Plus Ribavirin (N=312) | Peginterferon Alfa-2b Plus Ribavirin (N=286)
Gallstones (Hepatobiliary disorders) | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thoracic pain (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropaenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropaenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopaenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cryoglobulinaemia (Immune system disorders) | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0
Appendicitis (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Cell tissue inflammation (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vocal cord neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional Interferon Plus Ribavirin (N=62) | Peginterferon Alfa-2a Plus Ribavirin (N=312) | Peginterferon Alfa-2b Plus Ribavirin (N=286)
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 28 | 26
Itch (Skin and subcutaneous tissue disorders) | 9 | 50 | 44
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 16 | 16
Pain in extremities (Musculoskeletal and connective tissue disorders) | 1 | 15 | 16
Dorsalgia (Musculoskeletal and connective tissue disorders) | 1 | 9 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 51 | 33
Decreased appetite (Metabolism and nutrition disorders) | 12 | 75 | 52
Cachexia (Metabolism and nutrition disorders) | 2 | 9 | 17
Anaemia (Blood and lymphatic system disorders) | 11 | 109 | 111
Leucopaenia (Blood and lymphatic system disorders) | 1 | 14 | 20
Neutropaenia (Blood and lymphatic system disorders) | 3 | 60 | 45
Thrombocytopaenia (Blood and lymphatic system disorders) | 3 | 27 | 21
Headache (Nervous system disorders) | 19 | 67 | 67
Insomnia (Nervous system disorders) | 6 | 43 | 30
Dizziness (Nervous system disorders) | 5 | 28 | 25
Diarrhoea (Gastrointestinal disorders) | 3 | 21 | 27
Abdominal pain (Gastrointestinal disorders) | 1 | 10 | 16
High abdominal pain (Gastrointestinal disorders) | 7 | 25 | 23
Nausea (Gastrointestinal disorders) | 10 | 57 | 45
Vomiting (Gastrointestinal disorders) | 7 | 21 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 23 | 11
Anxiety (Psychiatric disorders) | 2 | 12 | 19
Depression (Psychiatric disorders) | 2 | 36 | 35
Irritability (Psychiatric disorders) | 4 | 41 | 31
Asthenia (General disorders) | 23 | 114 | 107
Pain (General disorders) | 3 | 19 | 30
Flu condition (General disorders) | 3 | 25 | 50
Fatigue (General disorders) | 9 | 36 | 35
Malaise (General disorders) | 7 | 19 | 21
Pyrexia (General disorders) | 16 | 65 | 66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.